CLINICAL TRIAL: NCT05715827
Title: A Prospective, Single-center, Single-arm, Pivotal Trial to Evaluate Safety and Efficacy of the Medtronic Hugo™ Robotic Assisted Surgery (RAS) System (Hello Hugo)
Brief Title: A Prospective, Single-center, Single-arm, Pivotal Trial of the Medtronic Hugo™ Robotic Assisted Surgery (RAS) System
Status: Completed | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT21028
Record Dates: First submitted 2023-01-27; First posted 2023-02-08 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer; Cholelithiases; Cholecystitis; Gallbladder Polyp
MeSH Terms: conditions — Prostatic Neoplasms; Cholelithiasis; Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Robotic Assisted Surgery (RAS) (Experimental): Robotic Assisted radical prostatectomy and cholecystectomy
  Interventions: Device: RAS prostatectomy and RAS cholecystectomy

INTERVENTIONS:
Device: RAS prostatectomy and RAS cholecystectomy — There are two types of interventions in the study.
  Patients indicated for Robotic Assisted Surgery (RAS) for a prostatectomy will have the RAS surgery using the Medtronic Hugo RAS system.
  Patients indicated for Robotic Assisted Surgery (RAS) for a cholecystectomy will have the RAS surgery using the Medtronic Hugo RAS system.

SUMMARY:
The goal of this clinical trial is to test the safety and effectiveness of the Medtronic Hugo™ RAS System in patients undergoing a prostatectomy or a cholecystectomy. A minimum of 40 subjects will be enrolled at single site in Republic of Korea: 20 for prostatectomy and 20 for cholecystectomy. All participants will be followed for 30 days (±7 days) post-procedure.

DETAILED DESCRIPTION:
This study is a prospective, single-center, single-arm, pivotal trial in 40 patients undergoing prostatectomy (N=20) or cholecystectomy (N=20) using the Medtronic Hugo™ RAS System.

The objectives of this study are:

* to confirm that the Medtronic Hugo™ RAS System performs as intended when used for prostatectomy or cholecystectomy
* to assess the short-term safety outcome of the Medtronic Hugo™ RAS System when used for prostatectomy or cholecystectomy

The Medtronic Hugo™ RAS System is intended to be used in this study for prostatectomy and cholecystectomy to be performed in subjects that meet the eligibility criteria. The subjects must be acceptable candidates for a fully robotic assisted procedure with the Medtronic Hugo™ RAS System, as determined by the principal investigator. Adult subjects indicated for a radical prostatectomy for clinically localized prostate cancer, or a cholecystectomy for cholelithiasis, cholecystitis, or gallbladder polyps will be included in this study. The study consists of following study visits:

* Baseline: When a subject is consented, the principal investigator will review the subject's medical record and confirms if they meet all specified inclusion criteria and none of the exclusion criteria.
* Surgical Procedure: The subject will arrive for admission to the hospital and prepped for surgery. The subject will receive a robotic assisted prostatectomy or cholecystectomy per indication.
* Up to Discharge: The subject's condition will be closely monitored until discharge. Vital signs and laboratory test will be conducted. For prostatectomy subjects, pathological exam results will be also collected.
* Post-Operative Follow-Up: Prostatectomy subjects will be followed at 7-day, 14-day (±3 days), and 30-day (±7 days) post-operative outpatient visits. Cholecystectomy subjects will be followed at 30-day (±7 days) post-operative outpatient visit.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (22 years old or greater) who are willing to participate and provide informed consent
2. Subjects indicated for a radical prostatectomy or a cholecystectomy

   * Prostatectomy: Male patients requiring radical prostatectomy for clinically localized prostate cancer (* Clinically localized prostate cancer is defined as following: biopsy-proven prostate adenocarcinoma, clinical staged as T1-T2N0M0 upon standard imaging findings such as bone scan, MRI, or CT)
   * Cholecystectomy: Patients requiring cholecystectomy for cholelithiasis, cholecystitis, or gallbladder polyps (* For gallbladder polyps, only followings will be considered: gallbladder polyps ≥10 mm, enlarging polyps, or symptomatic gallbladder polyps)

Exclusion Criteria:

1. Patient with a considerable risk for laparoscopic surgery (e.g., severe cardiopulmonary diseases which contraindicated to general anesthesia, uncontrolled coagulopathy, etc.)
2. Patients requiring urgent surgery
3. Pregnant or lactating women
4. Patients with either of followings:

   * Prostatectomy: Metastatic prostate cancer or estimated life expectancy less than 10 years
   * Cholecystectomy: Severe liver cirrhosis (Child-Pugh class C) with portal hypertension, suspicion of gallbladder cancer
5. Previous abdominal surgery (open or laparoscopic) within 2 years before enrollment
6. Concurrent participation in another clinical study that may confound study results
7. Patient has a condition that could compromise study compliance (e.g., mentally incompetent, alcohol or drug abuse) as determined by the investigator
8. Subjects who are considered unsuitable to conduct the trial as determined by the investigator

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-12 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwon W, Jang JY, Jeong CW, Anselme S, Pradella F, Woods J. Cholecystectomy with the Hugo robotic-assisted surgery system: the first general surgery clinical study in Korea. Surg Endosc. 2025 Jan;39(1):171-179. doi: 10.1007/s00464-024-11334-4. Epub 2024 Oct 28. PMID 39466427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from February 12, 2023, to May 7th, 2023.
  Subjects were recruited at Seoul National University Hospital, a major hospital in Seoul, Korea.
  Enrollment involved 42 subjects, with 20 subjects indicated for robotic-assisted Prostatectomy and 22 subjects indicated for robotic-assisted Cholecystectomy.
Pre-assignment Details: After enrollment, two Cholecystectomy subjects exited the study before surgery due to a surgeon's decision and a console communication error.
  These two subjects did not undergo a procedure with the Hugo™ RAS System and were treated with laparoscopy as Standard-of-care treatment.
Groups:
- Robotic Assisted Radical Prostatectomy: Robotic-assisted Radical Prostatectomy Patients indicated for Robotic Assisted Surgery (RAS) for a Prostatectomy will have the RAS surgery using the Medtronic Hugo RAS system.
- Robotic-assisted Cholecystectomy: Robotic-assisted Cholecystectomy Patients indicated for Robotic Assisted Surgery (RAS) for a Cholecystectomy will have the RAS surgery using the Medtronic Hugo RAS system.
Period: Overall Study
Arm/Group | Robotic Assisted Radical Prostatectomy | Robotic-assisted Cholecystectomy
Started | 20 | 22
Completed | 20 | 20
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — console communication error | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full Analysis Set (FAS) used to evaluate the primary and secondary endpoints was defined as all enrolled subjects in whom a Hugo™ RAS procedure began. Therefore, the 2 cholecystectomy subjects who did not undergo a procedure with the Hugo™ RAS System and exited the study before surgery were excluded from the FAS.
Groups:
- Robotic Assisted Prostatectomy: The study population will consist of patients 22 years of age or older indicated for a robotic assisted prostatectomy with Hugo™ RAS.
- Robotic Assisted Cholecystectomy: The study population will consist of patients 22 years of age or older indicated for a robotic assisted cholecystectomy with Hugo™ RAS.
- Total: Total of all reporting groups
Arm/Group | Robotic Assisted Prostatectomy | Robotic Assisted Cholecystectomy | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [62 to 74] | 58 [51 to 65] | 63 [56 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 12 | 12
  Male | 20 | 8 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 20 | 20 | 40
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 24.7 [24 to 26] | 23.9 [22 to 27] | 24.6 [23 to 26]

OUTCOME MEASURES:

1. Primary Outcome: Completion Rate
Description: The primary endpoint of this study is the completion rate, which is defined as a proportion of subjects who completed the surgery without conversion due to system serious malfunction, and without any major complications within 24-hour post-surgery.
Time Frame: 24 hours
Population: For the analysis, we considered the Full Analysis Set (FAS), defined as all enrolled subjects who began the Hugo™ RAS procedure (first skin incision). Subjects who consented but did not reach the first incision were excluded. Those converted to open or conventional surgery, not due to the Hugo™ RAS System, were included in the safety and descriptive analyses but excluded from the primary endpoint analysis.
Measure: Count of Participants; unit: Participants
Groups:
- RAS Prostatectomy: 20 subjects who were indicated for robotic-assisted Prostatectomy received a surgery with the Hugo RAS System.
- RAS Cholecystectomy: 20 subjects indicated for robotic-assisted Cholecystectomy received surgery with the Hugo RAS system
Arm/Group | RAS Prostatectomy | RAS Cholecystectomy
Number analyzed (Participants) | 20 | 20
Participants | 20 | 19
Statistical Analysis 1: Comparison: RAS Prostatectomy vs RAS Cholecystectomy; The study aimed to confirm the Medtronic Hugo™ RAS System's performance for prostatectomy or cholecystectomy, targeting a 95% completion rate (no conversion due to system issues or major complications within 24 hours). The Full Analysis Set (FAS) included all subjects starting the procedure. Descriptive statistics and 95% confidence intervals were used to assess primary and secondary endpoints, confirming safety and effectiveness; Test type: Other — The study used descriptive statistics and 95% confidence intervals to summarize data. The sample size of 40 patients (20 per surgery type) was based on prior studies with 3% device malfunction and 0.9% failure-related conversion rates. The primary endpoint was the completion rate, defined as ≥95% without conversion due to system issues or major complications within 24 hours. The Full Analysis Set included all subjects who started the procedure. No interim analyses were planned; The study used descriptive statistics and confidence intervals, not hypothesis testing with p-values. The main goal was to confirm the completion rate met or exceeded 95% and present a 95% confidence interval; The main goal was to confirm the completion rate met or exceeded 95% with a 95% confidence interval; Completion rate = 97.5, 95% CI 2-sided [86.8 to 99.9] — Estimated Value of 97.5% is an overall completion rate; Descriptive Analysis was used

2. Secondary Outcome: Overall Complication Rate Through 30-day Post-surgery
Description: A proportion of subjects with any post-operative complication within 30-days post-surgery using the investigational device
Time Frame: 30 days
Population: subjects who were indicated for robotic-assisted Prostatectomy and Cholecystectomy who went under procedure with Hugo RAS System
Measure: Count of Participants; unit: Participants
Arm/Group | RAS Prostatectomy | RAS Cholecystectomy
Number analyzed (Participants) | 20 | 20
Participants | 5 | 3
Statistical Analysis 1: Comparison: RAS Prostatectomy vs RAS Cholecystectomy; The secondary objective is to assess the short-term safety outcome of the Medtronic Hugo™ RAS System when used for prostatectomy or cholecystectomy. Overall complication rate through 30-day post-surgery: A proportion of subjects with any postoperative complication within 30-days post-surgery using the investigational device; Test type: Other — Descriptive statistics will be used, presenting frequency, percentage, and 95% confidence intervals for each secondary endpoint: overall complication rate, major complication rate, readmission rate, reoperation rate, and Device Deficiencies (DD) rate through 30 days post-surgery. Secondary endpoints will be assessed overall and by surgery type (prostatectomy and cholecystectomy); Descriptive statistics and estimated rates were used. P-values were not calculated for secondary endpoints; Overall Complication Rate = 20, 95% CI 2-sided [9.1 to 35.6]

3. Secondary Outcome: Major Complication Rate Through 30-day Post-surgery
Description: This measure reports the proportion of subjects with post-operative complications classified as Grade 3 or higher by the Clavien-Dindo system within 30 days post-surgery. The Clavien-Dindo system classifies post-operative complications from Grade 1 (minor) to Grade 5 (death).
  Grade 1: Minor deviation, no intervention. Grade 2: Requires medication or transfusion. Grade 3: Requires surgical, endoscopic, or radiological intervention. Grade 4: Life-threatening, requires ICU. Grade 5: Death. Higher grades indicate worse outcomes, with Grade 3 or higher classified as "major complications."
Time Frame: 30 days
Population: subjects indicated for robotic-assisted Cholecystectomy received surgery with Hugo RAS System
Measure: Count of Participants; unit: Participants
Arm/Group | RAS Prostatectomy | RAS Cholecystectomy
Number analyzed (Participants) | 20 | 20
Participants | 0 | 2
Statistical Analysis 1: Comparison: RAS Prostatectomy vs RAS Cholecystectomy; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; Descriptive statistics and estimated rates were used. P-values were not calculated for secondary endpoints; Major complication rate = 5, 95% CI 2-sided [0.6 to 16.9]

4. Secondary Outcome: Readmission Rate Through 30-day Post-surgery
Description: A proportion of subjects hospitalized within 30 days post-surgery
Time Frame: 30 days
Population: subjects who were indicated for robotic-assisted Prostatectomy and Cholecystectomy underwent the procedure with Hugo RAS system
Measure: Count of Participants; unit: Participants
Arm/Group | RAS Prostatectomy | RAS Cholecystectomy
Number analyzed (Participants) | 20 | 20
Participants | 1 | 3
Statistical Analysis 1: Comparison: RAS Prostatectomy vs RAS Cholecystectomy; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; Descriptive statistics and estimated rates were used. P-values were not calculated for secondary endpoints; Readmission rate = 10, 95% CI 2-sided [2.8 to 23.7]

5. Secondary Outcome: Reoperation Rate Through 30-day Post-surgery
Description: A proportion of subjects go through reoperation for the same indication within 30 days post-surgery
Time Frame: 30 days
Population: subjects who were indicated for robotic-assisted Prostatectomy and Cholecystectomy who underwent procedure with hugo RAS system
Measure: Count of Participants; unit: Participants
Arm/Group | RAS Prostatectomy | RAS Cholecystectomy
Number analyzed (Participants) | 20 | 20
Participants | 0 | 0
Statistical Analysis 1: Comparison: RAS Prostatectomy vs RAS Cholecystectomy; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; Descriptive statistics and estimated rates were used. P-values were not calculated for secondary endpoints; Reoperation rate = 0.0

6. Secondary Outcome: Device Deficiency Rate
Description: A proportion of subjects with any device deficiency (DD) during robotic assisted surgery using the investigational device
Time Frame: Peri-operative
Population: subjects who were indicated for robotic-assisted Prostatectomy and Cholecystectomy received a surgery with the Hugo RAS System.
Measure: Count of Participants; unit: Participants
Arm/Group | RAS Prostatectomy | RAS Cholecystectomy
Number analyzed (Participants) | 20 | 20
Participants | 10 | 3
Statistical Analysis 1: Comparison: RAS Prostatectomy vs RAS Cholecystectomy; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; Descriptive statistics and estimated rates were used. P-values were not calculated for secondary endpoints; Device deficiency rate = 32.5, 95% CI 2-sided [18.6 to 49.1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the study duration, including the baseline period, surgical procedure, up to hospital discharge, and during the follow-up visits, which extended up to 30 days post-surgery.
Description: In this study, an adverse event (AE) is defined as any untoward medical occurrence in a subject, which does not necessarily have a causal relationship with the study device. A serious adverse event (SAE) is any AE that results in death, is life-threatening, requires hospitalization, results in disability or permanent damage, or necessitates intervention to prevent permanent impairment or damage.
Arm/Group | RAS Prostatectomy | RAS Cholecystectomy
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20 | 3/20
Other Adverse Events (participants affected / at risk) | 4/20 | 2/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAS Prostatectomy (N=20) | RAS Cholecystectomy (N=20)
Asthenia (General disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small Bowel Nos Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall hematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
biliary tract disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAS Prostatectomy (N=20) | RAS Cholecystectomy (N=20)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-abdominal hemmorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot publish or disclose study results until a multicenter publication is released. If not published within one year after study completion at all sites, the PI may then publish, subject to review. The PI must submit publications to Medtronic 60 days before submission for review. Medtronic can request removal of Confidential Information, corrections, and may delay publication by up to 90 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT05715827/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT05715827/SAP_001.pdf